CLINICAL TRIAL: NCT04922476
Title: Open Label Clinical Trial on the Efficacy of a Probiotic Strain of Bifidobacterium Longum 35624 (Alflorex®) in Functional Gastrointestinal Disorders (GFRS) in Children 8 to 18 Years of Age.
Brief Title: Effect of 35624® Alflorex® in Functional Gastrointestinal Disorders (FGIDs) in Children.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PrecisionBiotics Group Ltd. (Industry)
Collaborators: Instituto de Nutrición y Tecnología de los Alimentos (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBCT002A
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Functional Gastrointestinal Disorders; Functional Abdominal Pain
Keywords: Bifidobacterium longum 35624®; Probiotic; Food supplement; Alflorex®
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotic (Experimental): Alflorex® The participants consume one probiotic capsule a day for 12 weeks.
  Interventions: Dietary Supplement: Alflorex®

INTERVENTIONS:
Dietary Supplement: Alflorex® — Each probiotic capsule contains 1 x 10^9 CFU of B. longum 35624® and corn starch, hydroxypropyl methyl cellulose and magnesium stearate.

SUMMARY:
The aim of this study is to evaluate the effect of supplementation with Bifidobacterium longum 35624® Alflorex® on frequency and severity of symptoms of abdominal pain using an adapted Irritable Bowel Symptom Severity Scoring System (IBS-SSS) to accurately reflect the pediatric population using the aid of the validated Numeric Pain Rating Scale (NRS-II) in children with Functional Gastrointestinal Disorders (FGIDs).

DETAILED DESCRIPTION:
This is an open label study to assess the safety and effectiveness of Bifidobacterium longum 35624® Alflorex® when consumed once daily by children with Functional Gastrointestinal Disorders (FGIDs). The 12-week intervention study will be conducted in 63 non-coeliac children aged 8 to 18 years old with an FGID who experience at least two episodes of abdominal pain per week. The study will consist of 5 visits over a 14 week period commencing with a screening visit. The second visit will be the baseline (start of intervention), followed by third (mid-intervention), fourth (end of treatment) and fifth (follow up) visit. Questionnaires will be administered from the second to the fifth visit. A blood sample will be taken before treatment to rule out coeliac disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8-18 years
2. Any sex
3. ROME IV diagnostic criteria Pediatric functional digestive disorders: in children and adolescents. H2. Functional abdominal pain disorders H2a. Functional dyspepsia H2b. Irritable bowel syndrome H2d. Functional abdominal pain not otherwise specified H3. Functional defecation disorders H3a. Functional constipation H3b. Non-retentive fecal incontinence Meet the criteria during the last three months with the onset symptoms for at least six months before diagnosis
4. IBS rated moderate to severe according to GSRS-IBS score (Spanish / LA)
5. At least two episodes of abdominal pain per week
6. No consumption of probiotics at least two weeks before baseline measurements (but preferably four weeks);
7. Dad, Mom, or Guardian able to understand the protocol;
8. Be willing to maintain stable dietary habits throughout the study period;
9. Be able to communicate well with the Investigator, to understand and comply with the requirements of the study and be judged suitable for the study in the opinion of the Investigator;
10. Signature of Informed Consent.

Exclusion Criteria:

1. Children with systemic, organic or metabolic diseases, immunosuppression, different from IBS
2. Previous major abdominal surgery;
3. Consumption of proton pump inhibitors, H2 antagonists;
4. Consumption of probiotics in the two weeks before baseline measurements;
5. Are less than 8 or older than 18 years of age at the time of consent;
6. Subject who has been on antibiotics during the past 3 months;
7. Subjects who have not had at least two episodes of abdominal pain per week;
8. Subject with a malignant disease or any concomitant end-state organ disease and/or laboratory abnormalities considered by Investigators to be risky or that could interfere with data collection;
9. Subject who are coeliac or lactose intolerant;
10. Known allergy to any of the components of the test product;
11. Participation in a clinical study with an investigational product within 60 days before screening, or plans to participate in another study during the study period;
12. Subject has a history of non-compliance;
13. Use of dietary supplements or other fermented foods that contain live bacteria.
14. Pregnant or lactating females.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2023-03-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Change in IBS symptom severity assessed by an adapted Irritable Bowel Symptom Severity Scoring System (IBS-SSS) | Change from baseline, assessed at 6 and 12 weeks of supplement intake
  The IBS-SSS measures symptom severity in IBS patients and is a reliable and validated questionnaire taking into account the composite score of abdominal pain, number of days with abdominal pain, bloating/distention, satisfaction with bowel habits and IBS-related quality of life. For this study, an adapted version was used in conjunction with the NRS-11 pain scale for the purposes of accurately capturing the response of a pediatric population. The NRS-11 pain scale goes from 0-10 with 0 indicating "no pain" and 10 indicating "very severe pain."
Change in abdominal pain assessed by the Numeric Rating Scale for pain | Change from baseline, assessed at 6 and 12 weeks of supplement intake
  The Numeric Rating Scale (NRS-11) is an 11-point scale for patient self-reporting of pain which goes from 0 (no pain) to 10 (worst pain)

SECONDARY OUTCOMES:
Change in quality of life assessed by the Irritable Bowel Syndrome-Quality of Life questionnaire | Change from baseline, assessed at 6 and 12 weeks of supplement intake
  The IBS-QOL scoring is from 0 to 100, with higher scores indicating better IBS specific quality of life
Change in stool consistency assessed using the Bristol Stool Form Scale | Change from baseline, assessed at 6 and 12 weeks of supplement intake
  The Bristol Stool Form Scale classifies stool according to shape and consistency and assigns a sample a number from 1-7 depending on its characteristics, corresponding to constipation normal or diarrhea.
Change in stool frequency | Change from baseline, assessed at 6 and 12 weeks of supplement intake
  Assessed from patient diaries
Change in days absent from school | Change from baseline, assessed at 6 and 12 weeks of supplement intake
  Assess from patient diaries

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Murphy, PhD, Study Director — PrecisionBiotics Group Ltd.
Locations (1):
- Instituto de Nutrición y Tecnología de los Alimentos, Universidad de Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No